CLINICAL TRIAL: NCT02205320
Title: A Comparative, Crossover, Pharmacokinetic, Pharmacodynamic and Safety Study of Three Forms of PEG-G-CSF in Normal Healthy Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PG-01-003
Record Dates: First submitted 2014-07-29; First posted 2014-07-31 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2014-07

CONDITIONS: Pharmacokinetics
Keywords: Pegfilgrastim; Pharmacokinetics; Pharmacodynamics; Healthy volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Treatment Sequence I (DRL, A, B) (Experimental): Patients will receive study drugs in the following cross-over sequence: DRL_PG, Pegfilgrastim Form A, Pegfilgrastim Form B. Each drug is administered as a single, 6 mg, subcutaneous injection.
  Interventions: Biological: DRL_PG; Biological: Pegfilgrastim Form A; Biological: Pegfilgrastim Form B
- Treatment Sequence II (DRL, B, A) (Experimental): Patients will receive study drugs in the following cross-over sequence: DRL_PG, Pegfilgrastim Form B, Pegfilgrastim Form A. Each drug is administered as a single, 6 mg, subcutaneous injection.
  Interventions: Biological: DRL_PG; Biological: Pegfilgrastim Form A; Biological: Pegfilgrastim Form B
- Treatment Sequence III (A, DRL, B) (Experimental): Patients will receive study drugs in the following cross-over sequence: Pegfilgrastim Form A, DRL_PG, Pegfilgrastim Form B. Each drug is administered as a single, 6 mg, subcutaneous injection.
  Interventions: Biological: DRL_PG; Biological: Pegfilgrastim Form A; Biological: Pegfilgrastim Form B
- Treatment Sequence IV (A, B, DRL) (Experimental): Patients will receive study drugs in the following cross-over sequence: Pegfilgrastim Form A, Pegfilgrastim Form B, DRL_PG. Each drug is administered as a single, 6 mg, subcutaneous injection.
  Interventions: Biological: DRL_PG; Biological: Pegfilgrastim Form A; Biological: Pegfilgrastim Form B
- Treatment Sequence V (B, A, DRL) (Experimental): Patients will receive study drugs in the following cross-over sequence: Pegfilgrastim Form B, Pegfilgrastim Form A, DRL_PG. Each drug is administered as a single, 6 mg, subcutaneous injection.
  Interventions: Biological: DRL_PG; Biological: Pegfilgrastim Form A; Biological: Pegfilgrastim Form B
- Treatment Sequence VI (B, DRL, A) (Experimental): Patients will receive study drugs in the following cross-over sequence: Pegfilgrastim Form B, DRL_PG, Pegfilgrastim Form A. Each drug is administered as a single, 6 mg, subcutaneous injection.
  Interventions: Biological: DRL_PG; Biological: Pegfilgrastim Form A; Biological: Pegfilgrastim Form B

INTERVENTIONS:
Biological: DRL_PG
Biological: Pegfilgrastim Form A
Biological: Pegfilgrastim Form B

SUMMARY:
This is a comparative pharmacokinetic, pharmacodynamic and safety study in healthy volunteers with three forms of pegylated granulocyte colony stimulating factors.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female subjects aged 18 to 55 years
2. A standardized body mass index
3. General good health as determined by the Investigator
4. Normal organ function as per the Investigator's judgement
5. Must be non-smokers, or ex-smokers who have not smoked within the previous 6 months from the screening visit
6. Female subjects must:

   * Not be lactating; not be pregnant
   * Agree to use an acceptable contraceptive method or be of non-childbearing potential
7. Male subjects must refrain from donating sperm or fathering a child during the study and until 3 months after the last study drug

Exclusion Criteria:

1. Known hypersensitivity to Escherichia coli derived proteins, pegfilgrastim, filgrastim or any other related component
2. Presence of antibodies to polyethylene glycol at screening
3. Positive result for cotinine (>500 ng/mL) or drugs of abuse at screening or on admission
4. Prior history of or current alcohol abuse or excessive intake of alcohol as judged by the Investigator
5. Donation of blood (≥500 mL) or plasma within the previous 3 months
6. History of unexplained syncopal episodes;
7. Any disorder that, in the Investigator's opinion, may interfere with study compliance
8. History of any cancer
9. History of pulmonary infiltrate or pneumonia within the previous 6 months from screening visit
10. Hereditary fructose and/or sorbitol intolerance
11. Absolute neutrophil count below 1500/mm3 or above 12000/mm3 at screening
12. Positive test for hepatitis B surface antigen, hepatitis C antibody, or human immunodeficiency virus (HIV) 1 or 2
13. Any abnormality in 12-lead ECG that in the Investigator's opinion is clinically significant and/or suggestive of underlying cardiac abnormalities
14. A clinical diagnosis of hypertension, significant hypercholesterolemia as judged by the Investigator, or thyroid abnormalities
15. Family history of acute myeloid leukemia or subjects with splenomegaly at baseline, or with sickle cell disease
16. Any prescribed or over the counter medications including analgesics, herbal remedies, vitamin therapy must not be used from 7 days prior to the first administration of study drugs

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 192 (Estimated)
Dates: Start 2014-02; Primary Completion 2014-08 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Cmax | 105 days
  Maximum plasma concentration
AUC(0-inf) | 105 days
  Area under concentration-time curve extrapolated from time 0 to infinity
AUC(0-t) | 105 days
  Area under concentration-time curve from time 0 to the time of the last quantifiable concentration
Emax | 105 days
  Maximum observed effect
AUEC(0-t) | 105 days
  Area under the effect time curve from time zero (predose) to last measured time

CONTACTS AND LOCATIONS:
Locations (1):
- QPS Bio-Kinetic, Springfield, Missouri, United States